CLINICAL TRIAL: NCT06881901
Title: Clopidogrel Monotherapy in Patients with Chronic Coronary Syndrome Following Coronary Artery Bypass Grafting : a Target Trial Emulation
Brief Title: Antiplatelet Strategy for CCS Patients Undergoing CABG
Acronym: CABG_DAPT_SAPT
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: Antiplatelet After CABG
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Coronary Syndrome; Coronary Artery Bypass Graft CABG
Keywords: antiplatelet drug; Dual antiplatelet therapy; Single antiplatelet therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dual antiplatelet therapy: Patients who were prescribed dual antiplatelet therapy (aspirin + clopidogrel) at the date of discharge from te index hospitalization for CABG
- Aspirin monotherapy: Patients who were prescribed single antiplatelet therapy (aspirin) at the date of discharge from te index hospitalization for CABG
- Clopidogrel monotherapy: Patients who were prescribed single antiplatelet therapy (clopidogrel) at the date of discharge from te index hospitalization for CABG

SUMMARY:
To evaluate the long-term outcomes of different antiplatelet strategies, including DAPT, aspirin monotherapy, and clopidogrel monotherapy, in CCS patients undergoing CABG. A retrospective, population-based cohort study was conducted using data from the Korean National Health Insurance Service (K-NHIS) database.

DETAILED DESCRIPTION:
The use of antiplatelet agents is crucial in preventing atherothrombotic complications and maintaining graft patency after coronary artery bypass grafting (CABG). While dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 inhibitor is recommended for one year in patients undergoing CABG for acute coronary syndrome (ACS), the optimal antiplatelet strategy for chronic coronary syndrome (CCS) remains unclear. In fact, current guidelines show discrepancies, with the American Heart Association/American College of Cardiology (AHA/ACC) recommending DAPT for one year to reduce the risk of saphenous vein graft (SVG) occlusion (Class IIb), while the European Society of Cardiology (ESC) recommends switching to aspirin monotherapy to reduce bleeding risk and considers DAPT only for high-risk patients (Class IIb). However, aspirin monotherapy may also not be the optimal alternative due to its limited efficacy in preventing thrombotic events and its inability to significantly reduce major bleeding compared to DAPT. Recently, clopidogrel monotherapy has emerged as a promising alternative, potentially offering both ischemic protection and a lower bleeding risk compared to DAPT even compared to aspirin monotherapy. An observational study comparing clopidogrel monotherapy with clopidogrel plus aspirin after CABG found that clopidogrel monotherapy demonstrated comparable to the combination therapy group. While this suggests that clopidogrel monotherapy could be a viable alternative, previous study was limited by its short follow-up duration and lack of bleeding outcome assessment. Thus, the investigators performed target trial emulation to evaluate long-term ischemic and bleeding outcomes associated with DAPT, aspirin monotherapy, and clopidogrel monotherapy in CCS patients following CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with underwent Coronary artery bypass surgery (CABG) between January 2010 and December 2020

Exclusion Criteria:

* In-hospital death
* Not prescribed SAPT or DAPT
* Received CABG due to myocardial infarction or had myocardial infarction
* Received CABG due to unstable angina or had unstable angina
* History of PCI
* Pre-existing Intracranial hemorrhage or gastrointestinal bleeding
* Oral anticoagulant prescription at discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were prescribed antiplatete therapy after undergoing CABG
Sampling Method: Non-Probability Sample
Enrollment: 29898 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 10 year after CABG
  Composite of all cause death, spontaneous MI, and stroke
Major GI bleeding | 10 year after CABG
  Major GI bleeding requiring transfusion

SECONDARY OUTCOMES:
All cause death | 10 year after CABG
  death from any cause
Spontaneous myocardial infarction | 10 year after CABG
  Myocardial infarction with hospitalozation
Stroke | 10 year after CABG
  Stroke after CABG
Repeat revascularization | 10 year after CABG
  Additional PCI or CABG after discharge
Bleeding evet | 10 year after CABG
  Any bleeding requiring transfusion

IPD SHARING:
Plan to Share IPD: No